CLINICAL TRIAL: NCT02034838
Title: Microboosting of Atazanavir 300 mg With 50 mg Versus 100 mg Ritonavir Daily in HIV-infected Patients: a Pharmacokinetic Study
Brief Title: Microboosting of Atazanavir 300 mg With 50 mg Versus 100mg Ritonavir Daily in HIV-infected Patients: a Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AI424-979; 20130609-01H (Other: Ottawa Hospital Research Institute)
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: HIV Infection
Keywords: PK; pharmacokinetic; HIV-infected; atazanavir; ritonavir
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- atazanavir 300mg boosted with ritonavir 100mg (Experimental): Two period drug interaction. Period one: atazanavir 300mg boosted with ritonavir 100 mg once daily as part of current treatment standard of care.
  Period two: atazanavir 300 mg boosted with ritonavir 50 mg once daily for study days 2-8 inclusive
  Interventions: Drug: atazanavir 300mg boosted with ritonavir 50 mg

INTERVENTIONS:
Drug: atazanavir 300mg boosted with ritonavir 50 mg — atazanavir 300 mg with ritonavir 100 mg once a day at 8:00 am for study day 1 and 9.
  atazanavir 300 mg with ritonavir 50 mg once a day at 8:00 am for 7 consecutive days (study days 2-8)
  Other Names: Reyataz; ATV; Norvir; RTV

SUMMARY:
This is an open-label, single group study to determine the pharmacokinetic profile of atazanavir 300 mg daily boosted with ritonavir 100mg daily in HIV-infected patients over a period of 9 days.

Ritonavir and atazanavir are protease inhibitors used to treat HIV. However, ritonavir, when used at low doses (up to 100mg) does not have HIV activity, but will enhance (boost) the blood concentrations of other drugs like atazanavir.

Recently, a study showed that taking 50mg of ritonavir administered in an oral solution led to similar blood concentrations of atazanavir than when given with 100mg of ritonavir. Potential benefits associated with a lower dose of ritonavir may include a reduction of side effects such as upset stomach and an improvement in cholesterol level. This study will look at the amount of atazanavir into your blood when given with ritonavir in a tablet formulation at 50mg or 100mg with standard atazanavir dose (300mg).

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the following criteria will be eligible for participation in this study:

  1. Signed informed consent prior to any study-related activities.
  2. Documented HIV infection.
  3. Male or female patients between 18 and 70 years of age inclusively.
  4. Medication history, vital signs and physical exam adequately showing no signs of acute illness at screening, as per the assessment by the physician.
  5. Patients must be willing to stop using any herbal or natural health products for 4 weeks prior to and during the study including:

     * Grapefruit, grapefruit juice, St. John's Wort and any others as determined by the investigators.
  6. Patients must be on an antiretroviral regimen with atazanavir/ ritonavir 300/100 mg daily as the only protease inhibitor plus any combination of nucleoside reverse transcriptase inhibitors, for at least four weeks.
  7. VL<40 copies/mL on the most recent measurement, during treatment with atazanavir 300 mg daily and ritonavir 100 mg daily, which must be within 12 weeks of the study start date.
  8. Reproductive Status: Definition of Women of Child-Bearing Potential (WOCBP). WOCBP comprises women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who are not post-menopausal (see definition below).

     * WOCBP must be using an acceptable method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of study drug in such a manner that the risk of pregnancy is minimized.
     * WOCBP must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent units of HCG) within 0 to 72 hours before the first dose of study drug.
     * Women must not be breast-feeding.
     * Sexually active fertile men must use effective birth control if their partners are WOCBP

Exclusion Criteria:

Patients meeting one or more of the following criteria will be excluded from the study:

1. Female patients of childbearing potential who:

   1. Has a positive urine pregnancy test at screening.
   2. Have not been using a barrier method of contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), for at least 3 months prior to participation in the study.
   3. Is not willing or able to use a reliable method of barrier contraception during the study.
   4. Is breastfeeding.
2. Patients with prior history of treatment failure on a PI based regimen, or with genotypic evidence of resistance associated mutations to protease inhibitors.
3. Use of any medication listed in Appendix I within 4 weeks prior to screening.
4. Use of any over-the-counter or prescription medications in the two weeks prior to Day 1 of the study that may interfere with absorption, distribution, metabolism or excretion of the study medications.
5. Inability to adhere to protocol.
6. Patients may be excluded from the study for other reasons, at the investigator's discretion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 9 days
  main pharmacokinetic parameters of atazanavir: AUC0-24h, Cmax and Cmin.

SECONDARY OUTCOMES:
adverse events | 9 days
  the main pharmacokinetic parameters of ritonavir: AUC0-24h, Cmax and Cmin, , adverse events and preference, as reported by patients during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: William Cameron, MD, FRCPC, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada